## **Study Title:** Improving Accessibility and Personalization of Cognitive Remediation for Schizophrenia

Clinicaltrials.gov: NCT03576976

Statistical Analysis
Date of Approval: 5/24/2018

## Improving Accessibility and Personalization of Cognitive Remediation for Schizophrenia

Statistical analyses for this project will focus on the comparison of proximal outcomes between Clinic and Hybrid delivery methods of Cognitive Remediation. There are two proximal outcomes: Treatment Satisfaction (primary) and Neurocognition (secondary).

Wilcoxon's rank sum test will be used to compare Clinic and Hybrid CR groups on treatment satisfaction at post-treatment and change on the average neurocognitive T score from baseline to post-treatment.